CLINICAL TRIAL: NCT02460146
Title: A Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Sequential Multiple Ascending, Repeat Doses of Oral CXA-10 in Healthy Obese Male Subjects
Brief Title: PK and PD of Sequential Multiple Ascending, Repeat Doses of Oral CXA-10 in Healthy Obese Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Complexa, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CXA-10-202
Record Dates: First submitted 2015-05-03; First posted 2015-06-02 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2016-05

CONDITIONS: Acute Kidney Injury
MeSH Terms: conditions — Acute Kidney Injury | interventions — CXA-10

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CXA-10 (Active Comparator): CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitrated oleic acid
  Interventions: Drug: CXA-10
- CXA-10 placebo (Placebo Comparator): The placebo contains olive oil with BHT (0.08% to 0.10%).
  Interventions: Other: CXA-10 placebo

INTERVENTIONS:
Drug: CXA-10 — CXA-10 (10-nitro-9(E)-octadec-9-enoic acid) is a specific isomer of nitrated oleic acid
  Arms: CXA-10
Other: CXA-10 placebo — The placebo contains olive oil with BHT (0.08% to 0.10%).
  Arms: CXA-10 placebo

SUMMARY:
The main purpose of this trial is to demonstrate the safety, tolerability and pharmacokinetics (PK) of CXA-10 and its metabolite(s) administered as multiple ascending oral doses over 14 days to healthy obese male volunteers.

DETAILED DESCRIPTION:
Complexa has developed an oral formulation of CXA-10. The main purpose of this trial is to demonstrate the safety, tolerability and pharmacokinetics (PK) of CXA-10 and its metabolite(s) administered as multiple ascending oral doses over 14 days to healthy obese male volunteers. The pharmacodynamic (PD) effects of CXA-10 on serum biomarkers, some of which are elevated in the obese population, will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >27 and ≤40 kg/m2
* In good general health as determined by a thorough medical history and physical examination, ECG, vital signs, and clinical laboratory evaluation
* Results of clinical laboratory tests must be without clinically significant abnormalities for this population and may exceed the limits of the reference ranges, including hematology, clinical chemistry and urinalysis except as noted below
* Hemoglobin A1c (HbA1c) <7%
* Average blood pressure <160/100 mmHg at screening
* QTcF interval (Fredericia's correction factor) must be ≤430 msec at screening and pre-dose

Exclusion Criteria:

* Any clinically relevant abnormality for this population identified on the screening history, physical or laboratory examinations, or any other medical condition or circumstance making the volunteer unsuitable for participation in the study
* Any clinical history of cardiovascular events, arrhythmias, fainting, palpitations, personal or family history of congenital prolonged QT syndromes or sudden unexpected death due to a cardiac reason
* History of any primary malignancy, including a history of melanoma or suspicious undiagnosed skin lesions, with the exception of basal cell or squamous cell carcinomas of the skin or cervical carcinoma in situ or other malignancies curatively treated and with no evidence of disease for at least 5 years
* History of regular alcohol consumption exceeding 21 units/week (one unit = 125 mL of wine or 284 mL of beer or a single 25 mL measure of spirits) within 6 months of screening
* Treatment with any prescription or non-prescription drugs (including vitamins, herbal and dietary supplements) within 7 days or 5 half-lives, whichever is longer, prior to dosing and until collection of the final PK sample. Use of any drug including aspirin or non-steroidal anti-inflammatory drugs (NSAIDs) must be avoided within 7 days prior to the first dose and during this study as it may interfere with the pharmacology of CXA-10. Use of high energy supplements or drinks (especially, those containing caffeine, protein supplements, and weight loss drugs)
* History of smoking, including e-cigarettes, or use of nicotine-containing products within 1 month of screening
* Resting heart rate ≥100 BPM after 5 minutes rest (as above) at the screening visit
* Subjects with any other clinically relevant ECG parameter abnormality (e.g., PR interval, QRS deviation) or any clinically significant ECG abnormality will be excluded from the study
* Any clinically significant murmurs evident on auscultation of the heart (including evidence of mitral valve prolapse)

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Safety (adverse events) and tolerability of multiple ascending oral doses of CXA 10 administered daily for 14 days | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Blok, MD, Principal Investigator — Jasper Clinic, Michigan
Locations (1):
- Jasper Clinical Research & Development, Inc., Kalamazoo, Michigan, United States

IPD SHARING:
Plan to Share IPD: No